CLINICAL TRIAL: NCT03689673
Title: A Prospective, Multicenter, Non-interventional Study to Describe the Effectiveness of Etiasa® (Sustained Release Granules of Mesalazine or 5-Aminosalicylate, or 5-ASA) in Maintenance Treatment of Ulcerative Colitis (UC )
Brief Title: Study of the Effectiveness of ETIASA® (Sustained Release 5-Aminosalicylate) in Maintenance Treatment of Ulcerative Colitis (UC)
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-58216-001
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection

SUMMARY:
The purpose of the protocol is to assess the effectiveness of Etiasa® for preventing relapse in Chinese patients with quiescent UC.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patient ≥ 18 years old and ≤ 65 years old
* Patient has provided written informed consent to participate in the study after the purpose and nature have been clearly explained to him/her;
* Patient with documented diagnosis of mild-moderate Ulcerative Colitis (UC). The "documented diagnosis" should include a typical histology observed at least once in the course of the disease;
* Have a documented history of UC that has been successfully maintained in complete steroid-free remission for at least 1 month prior to study entry;
* The modified mayo score ≤ 2, without subscore >1, which is supported by a rectum-sigmoidoscopy or a colonoscopy;
* Regimen of maintenance of remission contains Etiasa®
* Patient mentally and physically able to answer the questionnaire.

Exclusion Criteria:

* Have a history of allergy or hypersensitivity to salicylates, 5-aminosalicylates, or any component of Etiasa®;
* Pregnant and breastfeeding women, approaching childbirth female or unwilling to take birth control measures during the study;
* A topical 5-aminosalicylate agent is included in the regimen;
* Patients with infectious colitis (positive for germs, ovum or parasites causing bowel disease);
* Treated with the other study drug at enrollment, or within past 3 months of enrollment;
* Serious underlying disease other than UC which in the opinion of the investigator may interfere with the patient's ability to participate fully in the study;
* Crohn's disease;
* Pancreatitis;
* Known bleeding disorders;
* Potentially unreliable patients, and those judged by the investigator to be unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Median time to relapse according to the patients with different maintenance Etiasa® daily dose | Until relapse or maximum 5 years

SECONDARY OUTCOMES:
Relapse rates at 5 years or at study termination according to different maintenance Etiasa® daily dose | 5 years or at study termination
Calprotectin change from baseline to each hospital visit and relapse | From baseline up to 5 years
Hemoglobin change from baseline to each hospital visit and relapse | From baseline up to 5 years
C-reactive protein (CRP) change from baseline to each hospital visit and relapse | From baseline up to 5 years
Erythrocyte sedimentation rate (ESR) change from baseline to each hospital visit and relapse | From baseline up to 5 years
Interleukin-6 (IL-6) change from baseline to each hospital visit and relapse | From baseline up to 5 years
Colorectal cancer (CRC) incidence rate | Until relapse or maximum 5 years
Quality of Life (QoL) changes during the treatment | From baseline until relapse or 5 years or early termination
  Assessed by Inflammatory Bowel Disease Questionnaire (IBDQ) a health-related quality of life (HRQoL) tool measuring physical, social, and emotional status (score 10-70, poor to good HRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (26):
- China (26):
  - The Affiliated Beijing Chao-yang Hospital of Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - China-Japan Union Hospital of Jilin University, Changchun
  - The Third Affiliated Hospital of The Third Military Medical University of Chinese PLA, Chongqing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The First Affiliated Hospital of Sun Yatsen University, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yatsen University, Guangzhou
  - Hebi People Hospital, Hebi
  - Anhui Provincial Hospital, Hefei
  - Henan Province People Hospital, Henan
  - The PLA 150 Central Hospital, Luoyang
  - The First Affiliated hospital of Nan Chang University, Nanchang
  - Nanjing General Hospital of Nanjing Military Command, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Jiangsu Province Hospital of TCM, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Qingdao Municipal Hospital, Qingdao
  - Suzhou Third People Hospital, Suzhou
  - The second affiliated hospital of Suzhou University, Suzhou
  - Tianjin People's Hospital, Tianjin
  - The Second Hospital Affiliated to Wenzhou Medical College, Wenzhou
  - Union Hospital Affiliated to Tongji Medical College, Wuhan
  - The People's Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of the Fourth Military Medical University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou